CLINICAL TRIAL: NCT01663519
Title: Effectiveness of Insoles Provided to Diabetic Patients at Risk to Develop Ulcers
Brief Title: Effectiveness of Insoles Provided to Patients With Diabetes. A Longitudinal Randomized Controlled Study in Gothenburg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Hellstrand Tang, Certified Prosthetist & Orthotist, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VGFOUGSB-9725 Regional R&D
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Foot; Neuropathy; Quality of Life
Keywords: Diabetic foot; Offloading; Prevention; Orthotics
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prefabricated insoles (Experimental): Prefabricated insoles with support in medial arch and metatarsal pad. A 2 mm top layer of cushioned material.
  Interventions: Other: Prefabricated insoles
- Custom made insoles 35 shore (Experimental): Custom made insoles formed over an individual cast positive. 35 shore of hardness in material Ethyl Vinyl Acetate
  Interventions: Other: Custom made insoles 35 shore
- 55 shore Custom made insoles (Experimental): Custom made insoles formed over an individual cast positive. 55 shore of hardness in material Ethyl Vinyl Acetate
  Interventions: Other: 55 shore Custom made insole

INTERVENTIONS:
Other: Custom made insoles 35 shore — Insoles in Ethyl Vinyl Acetate (EVA) manufactured over an individual positive cast.
  Arms: Custom made insoles 35 shore
Other: Prefabricated insoles — Prefabricated insoles
  Other Names: Bauerfeind GloboTec® 312750501400
  Arms: Prefabricated insoles
Other: 55 shore Custom made insole — Insoles in Ethyl Vinyl Acetate (EVA) manufactured over an individual positive cast.
  Arms: 55 shore Custom made insoles

SUMMARY:
Introduction: Insoles and shoes are frequently prescribed to prevent foot ulcers in patients at risk of diabetes. A combination of neuropathy and foot deformities raises the risk from 1% to between 4-7% according to the Swedish National Board of Health and Welfare, Guidelines Diabetes Care 2010. Preventative care, which includes foot care, annual inspection of the feet, education and prescription of insoles in combination with well fitting shoes are supposed to decrease the risk of ulcers and prevent amputation. Further research is, however, needed to evaluate the effectiveness of these commonly prescribed insoles. The aim of this study is to compare three different types of insoles with respect to pressure distribution. Every 6 months follow-up is assessed until 24 months is reached.

DETAILED DESCRIPTION:
Patients included in the study were randomized into 3 different groups. Group number 1 and 2 got custom made insoles out of EVA (Ethyl Vinyl Acetate) with different hardness 35 and 55 shore respectively. Group nr 3 got prefabricated insole with support of the medial arch and in the forefoot. The top layer was covered with a 2 mm cushioned material, 25 shore, made out of microcellular urethane. All patients were recommended to wear good walking shoes with a semi rigid outer sole and stable heel counter. One and the same technician made the casting and fabricated the insoles as well as delivered the devices. Deliverance occured 2-3 weeks after the first visit.

At deliverance base line measurement was assessed.

ELIGIBILITY:
Inclusion criteria:

* First time visitor to Dept of Prosthetics & Orthotics
* Diabetes
* Age > 18 year
* Be able to walk independently
* Be able to read and understand Swedish

Exclusion Criteria:

* Ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-01; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
In shoe plantar pressure measurement | up to 24 months

SECONDARY OUTCOMES:
Gait analysis | every 6 months until 24 months is reached
  Optical tracking system with skin-mounted markers

OTHER OUTCOMES:
Health related quality of life | every 6 months until 24 months is reached
Cost and cost analysis | 24 month
  Calculation of costs for orthopaedic appliance in studied population

CONTACTS AND LOCATIONS:
Overall Officials: Roy Tranberg, PhD, Study Chair — Lundbergs laboratory for Orthopaedic Research
Locations (1):
- Lundbergs Laboratory for Orthopaedic Research, Gothenburg, Sweden

REFERENCES:
- [Result] Hellstrand Tang U, Zugner R, Lisovskaja V, Karlsson J, Hagberg K, Tranberg R. Comparison of plantar pressure in three types of insole given to patients with diabetes at risk of developing foot ulcers - A two-year, randomized trial. J Clin Transl Endocrinol. 2014 Jul 24;1(4):121-132. doi: 10.1016/j.jcte.2014.06.002. eCollection 2014 Dec. PMID 29159093
- [Result] Tang UH, Zugner R, Lisovskaja V, Karlsson J, Hagberg K, Tranberg R. Foot deformities, function in the lower extremities, and plantar pressure in patients with diabetes at high risk to develop foot ulcers. Diabet Foot Ankle. 2015 Jun 17;6:27593. doi: 10.3402/dfa.v6.27593. eCollection 2015. PMID 26087865
- See also: The Diabetic Foot - assessment and assistive devices — http://hdl.handle.net/2077/50860